CLINICAL TRIAL: NCT01085175
Title: A Multicenter, Phase II, Open Label Trial to Determine Optimal Imaging Parameters and Assess the Safety of LMI 1195 in Low Risk Patients and Heart Failure Patients With a History of Firing of an Implantable Cardioverter-Defibrillator
Brief Title: Trial to Determine Imaging Parameters of LMI1195 in Heart Failure Patients at Low and High Risk of Defibrillator Firing
Acronym: LMI1195-201
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor is re-evaluating the clinical development path
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LMI 1195-201
Record Dates: First submitted 2010-02-12; First posted 2010-03-11 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2011-02

CONDITIONS: Heart Failure
Keywords: Heart Failure,; PET Imaging,; Implantable Cardioverter-Defibrillator,; Sudden Cardiac Death
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Low risk Heart Failure patients
  Interventions: Drug: LMI 1195
- Cohort 2 (Experimental): High risk Heart Failure patients with history of Implantable Cardioverter-Defibrillator firing
  Interventions: Drug: LMI 1195

INTERVENTIONS:
Drug: LMI 1195 — Single bolus intravenous injection of LMI 1195
  Other Names: LMI 1195-101 Clinical Trial

SUMMARY:
The purpose of this clinical study is to determine the optimal imaging parameters and assess the safety of LMI1195 -101 in Heart Failure subjects at Low and High Risk of cardiac events.

DETAILED DESCRIPTION:
* To determine the optimal imaging protocol for a single dose of LMI1195 during positron emission tomography (PET) for the intended study population.
* To assess the safety and tolerability of LMI1195 in patients at low risk of ventricular arrhythmia ("low risk patients") and heart failure patients with a history of firing of an implantable cardioverter defibrillator (ICD) within 6 months prior to enrollment, a documented ejection fraction (EF) ≤ 35%, and a prior diagnosis of NYHA Class II-III heart failure ("heart failure patients") who are undergoing PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female ≥ 18 years of age
* a body weight that is <450 pounds
* Be able to lie flat for at least 2-hour intervals
* Have a normal left ventricular ejection fraction (i.e., ≥ 55% for cohort one or ≤35% for cohort two) by multiple gate acquisition scan (MUGA), echocardiogram or single photon emission computed tomography (SPECT) within 90 days prior, but no less than 3 days prior to enrollment.
* Have been scheduled to undergo or have undergone a SPECT or an approved PET perfusion imaging study performed within 90 days prior to, but no less than 3 days prior to enrollment. to and within the study timeline must be reviewed and deemed acceptable by the judgment of the investigator) (Additional More Specific Criteria can be accessed by contacting an LMI representative)

Exclusion Criteria:

* Have a history of diabetes, coronary artery disease, myocardial infarction heart arrhythmia (except sinus arrhythmia), heart failure, cardiomyopathy (e.g. restrictive, infiltrative or hypertrophic cardiomyopathy), constrictive pericarditis, myocarditis, complex congenital disease, surgically correctable valvular disease, and/or inoperable, obstructive valvular disease, pacemaker, syncope, transient ischemic attack (TIA) or cerebrovascular accident (CVA), Parkinson's disease, degenerative cerebral disease, or organ transplantation.significant comorbid conditions
* Have undergone major surgery within 4 weeks prior to enrollment or planned within 3 weeks after completion of the study.
* Unexplained syncope within 5 years.
* A life expectancy of < 1 year, from any cause.
* Are currently participating in another clinical trial of an investigational product.
* Have clinically significant laboratory abnormalities (e.g., liver enzymes, creatinine, etc.).
* Have a history of smoking within 1 month of enrollment.
* History of drug or alcohol abuse
* Have a history of major psychiatric disorder, active alcohol/drug abuse, and/or history of non-compliance.
* Receipt of any radiopharmaceutical within a period equal to 10 half-lives of the isotope (e.g., for 99mTc, a period of 60 hours; for 111In, a period of 28 days) prior to enrollment or receipt of any radiopharmaceutical containing iodine within a period of 3 months prior to enrollment.
* Have received any of the following medications within 30 days prior to enrollment, because of confounding effects to the autonomic nervous system: albuterol (Alupent, Ventolin within 24 hours), Dobutamine (Dobutrex), Dopamine (Intropin), Epinephrine (Adrenalin), Isoproterenol, Phenylephrine (Neo-Synephrine), Metaraminol (Aramine), Norepinephrine (Levophed), furazolidone (Furoxone), tricyclic antidepressants (Adapin, Asendin, Aventyl, Elavil, Endep, Norpramin, Pamelor, Sinequan, Surmontil, Tofranil, Vivactil), guanethidine (Ismelin), methyldopa (Aldomet). Over the counter herbs that have been reported to interact with adrenergic amines are excluded: ephedra (ma huang), St. John's wort; alfalfa; hibiscus; ginseng; angelica (dong quai); and yohimbe.
* Are not suitable subjects for completion of any screening or trial procedures including PET, scans & laboratory testing,
* Receipt of any radiopharmaceutical within a period of time that the agent has not decayed below background levels
* Have metal that cannot be removed from the body located in the thorax, Receiving Class I or III antiarrhythmic drug therapy, except for amiodarone.

(Additional More Specific Criteria can be accessed by contacting an LMI representative)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Dose acquisition time product, target and non-target F18 count density | Approximately one year

SECONDARY OUTCOMES:
Assess Image Quality Data Variability across age & sex stratification Determine Retention Index Values Determine Heart to Mediastinal Ratio Evaluate additional image derived markers that may have predictive value | Approximately one year

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Lee, M.D., Study Director — Lantheus Medical Imaging
Locations (1):
- Columbia University Medical College, New York, New York, United States